CLINICAL TRIAL: NCT00819546
Title: A Phase I Trial of Escalating Dose of RAD001 in Combination With PKC412 in Patients With Relapsed, Refractory or Poor Prognosis AML or MDS
Brief Title: RAD001 in Combination With PKC412 in Patients With Relapsed, Refractory or Poor Prognosis AML or MDS
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Richard Stone, MD (Other)
Collaborators: Beth Israel Deaconess Medical Center (Other); Massachusetts General Hospital (Other); Brigham and Women's Hospital (Other); Novartis (Industry)
Responsible Party: Sponsor-Investigator, Richard Stone, MD, Professor of Medicine, Dana-Farber Cancer Institute
Organization: Dana-Farber Cancer Institute (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 08-269
Record Dates: First submitted 2009-01-08; First posted 2009-01-09 (Estimated); Last update posted 2025-02-27 (Actual); Status verified 2025-02

CONDITIONS: Acute Myeloid Leukemia; Myelodysplastic Syndrome
Keywords: AML; MDS
MeSH Terms: conditions — Leukemia, Myeloid, Acute; Myelodysplastic Syndromes | interventions — Everolimus; midostaurin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Only one arm on this study. (Other)
  Interventions: Drug: RAD001; Drug: PKC412

INTERVENTIONS:
Drug: RAD001 — Participants will receive RAD001 on day 1 at the dose specified then again on days 8-28 for the first cycle. For all subsequent cycles RAD001 will be taken once daily.
  Other Names: everolimus
Drug: PKC412 — 50mg orally twice a day on days 2-28 for the first cycle. For all subsequent cycles 50mg of PKC412 will be taken orally twice daily.
  Other Names: midostaurin

SUMMARY:
The purpose of this research study is to determine the safety of the combination of RAD001 and PKC412 as a cancer treatment, and to establish the highest dose of RAD001 that can be given in conjunction with PKC412. These drugs have been used in other research trials for individuals with solid and hematology malignancies. Past research on PKC412 shows that it blocks the abnormal functioning of an enzyme called FLT3. FLT3 is found in your cells in either a normal (wild type) or genetically changed form and plays a role in the survival and growth of AML cells. RAD001 is an inhibitor of a central growth pathway that involves the protein MTOR. The MTOR pathway is overactive in cancer cells, causing the cells to grow abnormally. By inhibiting the abnormal growth activity of the MTOR pathway, RAD001 slows down and possibly stops the growth of cancer cells.

DETAILED DESCRIPTION:
* This is a dose-escalation study in which 3 participants will be given a particular starting dose of RAD001 on a certain schedule. If the dose and schedule are well tolerated, then the next 3 participants enrolled will be assigned a new dosing schedule and/or a higher dose of RAD001. This will continue until a maximum tolerated dose (MTD) is reached for RAD001.
* Each cycle of treatment consists of 28 days on an outpatient basis. Participants will receive RAD001 as the assigned schedule and dosage on day 1 and on days 8 through 28 for the first cycle. For all subsequent cycles RAD001 will be taken once daily. Additionally, all participants will take PKC412 twice a day on days 2 through 28 for the first cycle. For all subsequent cycles PKC412 will be taken twice daily.
* During the course of the trial the following evaluations and procedures will be completed at various times: review of medical history; review of concomitant medications; physical exam; performance status; vital signs; EKG; chest x-ray; blood tests and bone marrow aspirate/biopsy.

ELIGIBILITY:
Inclusion Criteria:

* Cytopathologically or histopathologically confirmed diagnosis of AML, MDS (RAEB-1, -2) or CMML, who are either relapsed or refractory to standard therapy, or are considered inappropriate candidates for standard therapy.
* Inappropriateness for standard therapy requires a) MDS patients: not be a candidate for immediate allogeneic stem cell transplantation, not have a -5q-cytogenetic abnormality (unless previously received lenalidomide), and not be an appropriate candidate for a DNA hypomethylating agent b) AML patients must be 60 years of age or greater and have one of more of the following documented poor risk factors: ECOG Performance Status = 2, 70 years of age or older, unfavorable cytogenetics.
* Life expectancy of at least 12 weeks
* Not likely to require cytoreductive therapy within one month (other than hydroxyurea)
* ECOG Performance Status of 2 or less
* Serum transaminase activity (AST/SGOT & ALT/SGPT) < 2.5 x ULN
* Serum total bilirubin < 1.5 x ULN ( with the exception of individuals with Gilbert's disease)
* INR < 1.3 (or < 3 on anticoagulants)
* Fasting serum cholesterol 300mg/dl or 7.75 mmol/L or less AND fasting triglycerides 2.5 ULN or less

Exclusion Criteria:

* Prior allogeneic, syngeneic, or autologous bone marrow transplant or stem cell transplant less than 2 months previously
* Female patients who are pregnant or breast feeding or adults of child bearing not employing double barrier contraception
* Concurrent severe and/or uncontrolled medical or psychiatric condition which may interfere with the completion of the study
* Impairment of gastrointestinal function or GI disease that may significantly alter absorption of PKC412 or RAD001
* Uncontrolled active infection
* Any pulmonary infiltrate on teh baseline chest x-ray known to be new in the previous 4 weeks
* Patients with a Grade 2 or higher hypercholesterolemia or hypertriglyceridemia despite lipid-lowering therapy
* Patients with history of another malignancy within the past 5 years, with the exception of adequately treated basal or squamous cell skin carcinoma or cervical carcinoma in situ
* History of non-compliance to medical regimens and patients who are unwilling or unable to comply with this protocol
* Prior treatment with any investigational drug within preceding 4 weeks
* Chronic treatment with systemic steroids or another immunosuppressive agent
* Patients should not receive immunization with attenuated live vaccines within one week of study entry or during study period
* Any severe or uncontrolled medical conditions or other conditions that could affect their participation
* Known history of HIV seropositivity
* Known hypersensitivity to RAD001 or other rapamycins or to its excipients
* Known hypersensitivity to PKC412 or to its excipients
* Diagnosis of acute promyelocytic leukemia

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 29 (Estimated)
Dates: Start 2009-01; Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
To identify the maximum tolerated dose of RAD001 that can be given in combination with twice daily PKC412 in patients who are non-chemotherapy candidates with AML or MDS. | 2 years

SECONDARY OUTCOMES:
To determine the toxicities of combination of RAD001 and PKC412. | 2 years
Observe anti-leukemic effects of this combination including a coda of patients with mutant FLT3 AML. | 2 years
Measure pharmacokinetics of each agent when administered in combination. | 2 years
Observe the pharmacodynamic effects on the phosphorylation of FLT3 and on activation of relevant signaling pathways and correlate such activation with response. | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Richard Stone, MD, Principal Investigator — Dana-Farber Cancer Institute
Locations (3):
- United States (3):
  - Massachusetts General Hospital, Boston, Massachusetts
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts